CLINICAL TRIAL: NCT04141267
Title: Feasibility of Isoflurane Sedation Using an Anesthetic-conserving Device in Prehospital Emergency Medicine: A Retrospective Study
Brief Title: Inhaled Sedation Using the Anesthetic-conserving Device ( ANACONDA) in Prehospital Emergency Medecine.
Acronym: ANACONDA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ANACONDA (29BRC19.0016)
Record Dates: First submitted 2019-08-06; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-02

CONDITIONS: Endotracheal Intubation; Deep Sedation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Achieving the optimal sedation level for patient management is not always possible using our standard intravenous medications in Pre-hospital Emergency medicine. Inhaled sedation is possible with the Anesthetic-conserving device with a standard respirator.

The pharmacodynamics and pharmacokinetics of halogenated agents allow deep sedation quickly after absorption.

The feasibility of inhaled sedation has never been studied in hospital.

DETAILED DESCRIPTION:
Retrospecive clinical monocentric study with sedated ventilated patients with isoflurane with the AnaConda® system out of hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient sedated by isoflurane with Anesthetic-conserving device in pre-hospital
* Major patient
* not opposed to participating

Exclusion Criteria:

* Adults Under legal protection
* patient refusal to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who were sedated by isoflurane with Anesthetic-conserving device in pre-hospital by the emergency teams of SAMU 29
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
depth of sedation | up to 1 day
  depth of sedation (measured by the Ramsay Score) 10 minutes from start of the sedation and at stop of pre hospital sedation. The Ramsay score ranges level of sedation from 1(patient anxious ,agitated,restless) to 6 (patient exhibits no response).

SECONDARY OUTCOMES:
hemodynamic tolerance of patients during isoflurane sedation | up to 1 day
  comparison of heart rate (heart beats per minute) before isoflurane start and 10 minutes from start of the sedation and at stop of pre hospital sedation
hemodynamic tolerance of patients during isoflurane sedation | up to 1day
  comparison of medium blood pressure (mmHg) before isoflurane start and 10 minutes from start of the sedation and at stop of pre hospital sedation

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie result in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three months and ending five years following the publication
Access Criteria: Data access requests will be rewiewed by internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.